CLINICAL TRIAL: NCT01406184
Title: RCT Evaluation of the Durham Connects Universal Newborn Nurse Home Visiting Program
Brief Title: Durham Connects RCT Evaluation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: The Duke Endowment (Other); The Pew Charitable Trusts (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00020974; Pro00017478 (Other: Duke University Health System Institutional Review Board); 1R01HD069981 (NIH); Pro00020974 (Other: Duke University Health System Institutional Review Board); Pro00027652 (Other: Duke University Health System Institutional Review Board)
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Unspecified Child Maltreatment, Suspected; Unspecified Child Maltreatment, Confirmed
Keywords: Child Abuse; Child Neglect; Child Hospital Emergency Room Presentations; Child Well-Care Compliance; Child Immunization Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Durham Connects Eligible Group (Experimental): From July 1, 2009 - December 31, 2010, all even-birth-date residential births in Durham County, North Carolina were randomly assigned to receive the Durham Connects nurse home visiting program.
  Interventions: Other: Durham Connects
- Control Group (No Intervention): From July 1, 2009 - December 31, 2010, all odd-birth-date residential births in Durham County, North Carolina were randomly assigned to a control group condition. These families were assigned to receive services as usual and served as the randomized comparison group for evaluating Durham Connects program impact.

INTERVENTIONS:
Other: Durham Connects — The program consists of 4-7 intervention contacts, including 1) a hospital birthing visit when a staff member schedules an initial home visit; 2) 1-3 nurse home visits between 3-12 weeks of infant age to provide physical assessments for infant and mother, intervention and education, assessment of family-specific needs, and connections to matched community resources, as needed, to provide longer-term support; 3) 1-2 nurse contacts with community service providers to facilitate successful connections; and 4) a telephone follow-up one month after case closure to review community connection outcomes. With family consent, letters from the program reporting on the visit are also provided to also connect families to maternal and infant healthcare providers for ongoing support.
  Arms: Durham Connects Eligible Group

SUMMARY:
The aim of this randomized controlled trial (RCT) is to evaluate the impact and mechanisms of the Durham Connects (DC) brief universal nurse home-visiting program to prevent child maltreatment and improve child well-being. It is the first-ever RCT of a home-visiting program that is designed to prevent child maltreatment in an entire community population.

Evaluation of program impact will test three hypotheses: 1) Random assignment to the Durham Connects Program will be associated with lower rates of child maltreatment and emergency department maltreatment-related injuries, better pediatric care, better parental functioning, and better child well-being than assignment as control; 2) Intervention effect sizes will be larger for higher-risk groups; and 3) Community resource use and enhanced family functioning will mediate the positive impact of Durham Connects on outcomes.

DETAILED DESCRIPTION:
The Durham Connects Program is an innovative, community based, universal nurse home-visiting program that aims to lower the population rate of child maltreatment and improve mother and child health and well-being. The Durham Connects Program is implemented jointly by the Durham County (North Carolina) Department of Public Health, the Center for Child & Family Health (a community non-profit), and Duke University. It is designed to be brief and inexpensive per family so that communities can afford its costs. Its goals are consistent with those of more intensive nurse home-visiting programs: 1) to connect with the mother in order to enhance maternal skills and self-efficacy; and 2) to connect the mother with needed community services such as health care, child care, mental health care, and financial and social support; so that 3) the mother can connect with her child.

DC achieves population reach by engaging all families within the community, rapidly triaging families based on identified risk to concentrate resources to families with greater needs, and connecting those families with significant nurse-identified risk to matched community programs and services to provide long-term support and a first step into the community system of care. The program consists of 4-7 manualized intervention contacts, including 1) a hospital birthing visit when a staff member communicates the importance of community support for parenting and schedules an initial home visit; 2) 1-3 nurse home visits between 3-12 weeks of infant age to provide physical assessments for infant and mother, intervention and education, assessment of family-specific needs, and for families with significant nurse-identified risk, connections to matched community resources to provide longer-term support; 3) 1-2 nurse contacts with community service providers to facilitate successful connections; and 4) a telephone follow-up one month after case closure to review consumer satisfaction and community connection outcomes. With family consent, letters from the program reporting on the visit are also provided to also connect families to maternal and infant healthcare providers for ongoing support.

During home visits, the nurse engages the mother (and father, when possible) to provide brief educational interventions for all families (e.g., safe sleep) and utilizes a high-inference approach to assess family needs across 12 empirically-derived factors linked to child health and well-being:

Healthcare: parent health, infant health, health care plans; Parenting/childcare: childcare plans, parent-infant relationship, management of infant crying; Family violence/safety: material supports, family violence, maltreatment history; and Parent well-being: depression/anxiety, substance abuse, social/emotional support.

The nurse scores each of the 12 factors and intervenes accordingly. A score of 1 (low risk) receives no subsequent intervention. A score of 2 (moderate risk) receives short-term, nurse-delivered intervention over 1-2 sessions. For a score of 3 (high risk) the nurse connects the family to matched community resources tailored to address that particular risk (such as, treatment for postpartum depression, a DSS social worker exclusively serving Durham Connects families for enrollment in Medicaid or food stamps, a multi-year home visiting program for long-term parent support). The nurse also provides follow up to make sure that each connection "sticks," requiring additional contacts with the family or community agency. A score of 4 (imminent risk) receives emergency intervention (<1% of cases). A final contact four weeks after case closure ascertains community connection outcomes and whether further problem solving is needed to address new or existing needs.

From July 1, 2009-December 31, 2010, all 4777 resident births from two Durham County hospitals (one academic tertiary care hospital and one community hospital) were randomized at the even-odd birth date group level, with families assigned to one of two intervention groups based on infant birth date: 1) even birth date families (n=2327) were randomly assigned to receive DC; DC staff attempted to schedule and visit all even birth date families; 2) odd birth date families (n=2450) were randomly assigned to receive other community services as usual and served as the control group. All eligible families (i.e., families living in Durham County giving birth at one of the two county hospitals) were included with experimental rigor, and without exception, but with ethical care for confidentiality. Hospital discharge records were utilized to confirm eligibility for all RCT families. The Duke University Health System Institutional Review Board approved all RCT implementation and evaluation procedures.

Completely independent of program implementation, a random, representative subsample of 549 families was selected to conduct an independent evaluation of DC beginning at infant age 6 months (initial interviews completed between infant ages 6-8 months). Use of random subsamples for evaluation of population-level interventions allows for testing of intervention impact while minimizing evaluation costs (e.g., Moving to Opportunity for Fair Housing intervention15). Consistent with this evaluation strategy, one family was randomly selected by computer algorithm from public birth records for each of the 549 days of the 18-month RCT enrollment period in order to examine program impact for families enrolled across the entire trial period. Families were selected from the entire population of eligible birth records (i.e., resident Durham County births at one of the two county birthing hospitals) without consideration for intervention participation or adherence. Selected families that declined participation were replaced with a randomly selected family with the same child birth date and race/ethnicity as the original family, in order to preserve any lack of selection bias based on these characteristics.

Selected families were contacted and invited to participate in a descriptive research study about family community service use and child development. Families were blind to study goals, and home interviewers were blind to family DC participation status. Overall, 682 families were randomly selected and 549 (81%) participated (n=269 DC-eligible families; n=280 control families). Post-hoc comparisons of hospital discharge records and public birth records after all evaluation study consenting and interviews were complete identified 18 participating families that were subsequently declared ineligible due to hospital discharge record error (n=13 families with no hospital discharge record; n=3 families with child birth date discrepancies; and n=2 families with address discrepancies affecting Durham County residency), resulting in a final sample of 664 selected families and 531 participating families. The ineligible families (n=9 DC-eligible families; n=9 control families) were removed without consideration for intervention adherence or evaluation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Infant born between July 1, 2009 and December 31, 2010
* Infant born at Durham County, North Carolina (NC) hospital (Duke or Durham Regional)
* Family of infant resides in Durham County, NC

Exclusion Criteria:

* Infant born before July 1, 2009 or after December 31, 2010
* Infant not born at Durham County, NC hospital
* Family of infant resides outside of Durham County, NC

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2329 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
DSS Investigated and Substantiated Child Maltreatment Rates | 0 - 12 Years of Child Age
  North Carolina Department of Social Services (DSS) reported lifetime cases of investigated and substantiated maltreatment caseness

SECONDARY OUTCOMES:
Child Emergency Room (ER) Presentation Rates | 0 - 12 Years of Child Age
  Lifetime child emergency department visits reported in hospital administrative records
Child Overnight Stays in Hospital | 0 - 12 Years Months of Child Age
  Lifetime child overnight stays in hospital for all overnight stays unrelated to the birthing stay as reported in hospital administrative records.
Child Postnatal Well-Care Compliance Rates | 0 - 24 Months of Child Age
  Rates of child compliance with well-care pediatric visits as reported by the mother
Child Social-Emotional Competence and Behavior Problems | 24 - 66 Months of Child Age
  Mothers complete the Head Start Competence Scale (Domitrovich et al., 2001), measuring child social and emotional skills central to interpersonal relationships and emotion regulation. Mothers also complete the ages 1.5-5 version of the Child Behavior Checklist (CBCL 1.5-5; Achenbach & Rescorla, 2001), a standardized measure assessing emotional and behavioral problems, including: 1) affective problems; 2) anxiety problems; 3) pervasive developmental problems; 4) Attention Deficit/Hyperactivity problems; and 5) Oppositional Defiant problems.
Mother Mental Health | 0-66 Months of Child Age
  Rates of mother depressive symptoms and anxiety symptoms as reported by the mother
Family Connections to Community Services/Resources | 0-66 Months of Child Age
  Rates of family connections to community resources and services as reported by the mother
Mother Parenting Behaviors | 0-66 Months of Child Age
  Rates of mother positive and negative parenting behaviors as reported by the mother or rated by an independent observer during in-home interviews or videotaped parent-child interactions

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Dodge, Ph.D., Principal Investigator — Duke University; Robert Murphy, Ph.D., Principal Investigator — Center for Child & Family Health; Karen O'Donnell, Ph.D., Principal Investigator — Center for Child & Family Health; W. Benjamin Goodman, Ph.D., Principal Investigator — Duke University
Locations (1):
- Center for Child and Family Policy, Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dodge KA, Goodman WB, Murphy RA, O'Donnell K, Sato J, Guptill S. Implementation and randomized controlled trial evaluation of universal postnatal nurse home visiting. Am J Public Health. 2014 Feb;104 Suppl 1(Suppl 1):S136-43. doi: 10.2105/AJPH.2013.301361. Epub 2013 Dec 19. PMID 24354833
- [Result] Dodge KA, Goodman WB, Murphy RA, O'Donnell K, Sato J. Randomized controlled trial of universal postnatal nurse home visiting: impact on emergency care. Pediatrics. 2013 Nov;132 Suppl 2(Suppl 2):S140-6. doi: 10.1542/peds.2013-1021M. PMID 24187116
- [Result] Dodge KA, Goodman WB, Murphy R, O'Donnell K, Sato J. Toward Population Impact from Home Visiting. Zero Three. 2013 Jan 1;33(3):17-23. PMID 23526864
- [Result] Alonso-Marsden S, Dodge KA, O'Donnell KJ, Murphy RA, Sato JM, Christopoulos C. Family risk as a predictor of initial engagement and follow-through in a universal nurse home visiting program to prevent child maltreatment. Child Abuse Negl. 2013 Aug;37(8):555-65. doi: 10.1016/j.chiabu.2013.03.012. Epub 2013 May 6. PMID 23660409
- [Result] Goodman WB, Dodge KA, Bai Y, O'Donnell KJ, Murphy RA. Randomized controlled trial of Family Connects: Effects on child emergency medical care from birth to 24 months. Dev Psychopathol. 2019 Dec;31(5):1863-1872. doi: 10.1017/S0954579419000889. PMID 31477190
- [Result] Goodman WB, Dodge KA, Bai Y, Murphy RA, O'Donnell K. Effect of a Universal Postpartum Nurse Home Visiting Program on Child Maltreatment and Emergency Medical Care at 5 Years of Age: A Randomized Clinical Trial. JAMA Netw Open. 2021 Jul 1;4(7):e2116024. doi: 10.1001/jamanetworkopen.2021.16024. PMID 34232300
- [Result] Dodge KA, Goodman WB, Bai Y, Best DL, Rehder P, Hill S. Impact of a universal perinatal home-visiting program on reduction in race disparities in maternal and child health: Two randomised controlled trials and a field quasi-experiment. Lancet Reg Health Am. 2022 Aug 23;15:100356. doi: 10.1016/j.lana.2022.100356. eCollection 2022 Nov. PMID 36778074
- [Result] Baziyants GA, Dodge KA, Bai Y, Goodman WB, O'Donnell K, Murphy RA. The effects of a universal short-term home visiting program: Two-year impact on parenting behavior and parent mental health. Child Abuse Negl. 2023 Jun;140:106140. doi: 10.1016/j.chiabu.2023.106140. Epub 2023 Mar 22. PMID 36963242
- See also: Center for Child & Family Policy, Duke University — http://childandfamilypolicy.duke.edu/
- See also: Center for Child & Family Health — http://www.ccfhnc.org/
- See also: Family Connects Website — http://www.familyconnects.org/

DOCUMENTS (1):
  • Informed Consent Form (2009-12-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT01406184/ICF_000.pdf